CLINICAL TRIAL: NCT02282540
Title: Novel Imaging of the Eustachian Tube; Patient Study
Acronym: CT-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Benedicte Falkenberg-Jensen, MD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ET31068
Record Dates: First submitted 2014-09-29; First posted 2014-11-04 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Otitis Media With Effusion; Eustachian Tube Disorder
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iodixanol to the Eustachian tube (Experimental): Iodixanol contrast medium diluted with NaCl to 20% into the tympanostomy tube while the patient lies on his / her back with the head slightly turned to the opposite side. After 10 minutes the CT examination will be conducted using 200 mA and 120 kV.
  Interventions: Procedure: Iodixanol to the Eustachian tube

INTERVENTIONS:
Procedure: Iodixanol to the Eustachian tube — Application of iodixanol to the middle ear for imaging of the ET.

SUMMARY:
The purpose of the study is to establish wether a contrast medium applied to the middle ear can be used to diagnose pathology in the auditory tube. We will examine patients with and without middle ear disease with CT after the application of an iodine based contrast medium.

DETAILED DESCRIPTION:
Introduction Dysfunction in the auditory tube / Eustachian tube (ET) is a frequent problem that may cause a series of middle ear conditions. Middle ear atelectasis, retraction of the tympanic membrane, in some cases "retraction pocket type-cholesteatoma" (5), chronic otitis, perforation of the tympanic membrane and conductive hearing loss due to poor middle ear ventilation are all associated with ET-dysfunction. The ET consists of two parts, the mobile cartilaginous part medially, and the fixated bony part laterally. The bony part is demarcated by thin bony walls and situated in the close proximity of vulnerable anatomical structures, while the cartilaginous part is supported by parapharyngeal soft tissue. Recent years, a new treatment procedure of ET balloon dilation has emerged. Restoration of ET function has offered a new approach for this large group of patients with great reduction of symptoms and secondary middle ear disease.

Only the cartilaginous part of the ET is accessible for treatment procedures. We also know that 20% of the patients dilated do not respond to dilation, and relapse of middle ear disease occurs (2). At present, no diagnostic procedure can distinguish between later responders and non-responders to dilation. Therefore, level diagnostics of obstruction and possibly identification of other discriminating parameters are important. Computer tomography (CT) is considered necessary before any type of tube intervention, mainly to exclude obstruction in the bony part of the tube or identification of any other pathoanatomical condition to contraindicate balloon dilatation. Visualisation of obstructions in the cartilaginous part is not possible with today's methods. Nor does the method provide any information on tube function.

There is a need for better diagnostic imaging of the ET. In this project we plan to develop a method for contrast medium application to the ET via the middle ear followed by CT imaging. The purpose is to tell whether the ET is open or on which level it is obstructed. So far some publications have showed that contrast media can pass through the ET (6,7,8), but no systematic trials have been published, clarifying the potential of the method.

We have recently conducted studies on temporal bone specimens from human cadavers and on 8 living rabbits. Results from these studies are not yet published, but our hypotheses are supported that the method for ET visualisation is feasible, safe, and that contrast media passes unhindered through a normal ET after application in the middle ear (6,7,8).

Hence the next step of the trial is to explore whether the method provides new information in human subjects with and without tube dysfunction.

Hypotheses Contrast medium applied in the middle ear passes through the ET and is visualised in the epipharynx in the following CT examination of the temporal bone in individuals with healthy middle ears and ET.

Contrast media applied in the middle ear does not pass through the entire ET and is not visualised in the epipharynx in the following CT examination of the temporal bone in individuals in the patient group.

It is possible to identify a highest level of obstruction after contrast media application in the middle ear based on visual identification of the lowest visible level of contrast medium in the ET in the following CT examination of the temporal bone in the patient group.

Level of obstruction of the ET predicts outcome of ET balloon dilation.

Material One fifth of chronic patients with otitis media with effusion (OME) have no beneficial effect of balloon dilation (2). We hypothesize that contrast media will not pass through the bony part of the ET in a majority of these patients, while it does in a majority of the patients experiencing successful relief of disease after balloon dilation. Variation is not known, but is presumed not to exceed 20%. Sample size calculation is not straight-forward in this case, handling dichotomous variables. Power calculation indicates a needed number of 80 individuals in the patient group to have a power of at least 80% for the detection of difference between these 2 groups with an alpha level of 5% with two-sided tests. Additionally, we include 15 controls with presumed healthy middle ears and ET to verify significantly better contrast media passage to epipharynx in these individuals than in the group of patients with chronic OME, based on similar power calculation.

Recruitment of this number to undergo a CT examination with contrast carefully administered through the tympanostomy tube will be done during a clinically indicated and planned CT to avoid excess radiation dose and additional visits to the hospital for the patients.

Mb Meniere patients are occasionally treated with tympanostomy tubes, although they do not have middle ear pathology. This patient group also routinely undergoes CT-examination of the temporal bone. Hence we plan to include 10 patients with mb Meniere and tympanostomy tubes to be examined with a similar contrast medium CT protocol as described above as a healthy control group.

Method Out patients referred to the Ear, nose and throat (ENT)-clinic for OME will be offered to be part of the study, given that they qualify according to the inclusion and exclusion criteria. All patients will be given written information and a consensus form.

At their first visit, the ENT- surgeon will control the status of the eardrum and middle ear by otomicroscopy. The extent of pneumatisation / atelectasis and fluid in the middle ear will be evaluated in addition to the state and position of the tympanic membrane. With a nasal endoscope the condition of Rosenmullers fossa and the function of torus tubarius will be examined. The latter is controlled by asking the patient to equalize pressure while the scope is in the nasopharynx, and the opening of the torus can be seen. The patients and controls are interviewed structurally for symptoms related to middle ear and temporal bone disease.

Included patients without a tympanostomy tube will be given one the same day as the clinical examination. The patients who are not treated with nasal corticosteroids will be prescribed them for use up until the first control.

CT will be performed after 3-4 weeks. At the CT-lab an ENT-surgeon will drip 2 ml iodixanol contrast medium diluted with saline (NaCl) to 20% into the tympanostomy tube while the patient lies on his / her back with the head slightly turned to the opposite side. After turning the head to a neutral position and a delay of 10 minutes the CT examination will be conducted using 200 milliampere (mA) and 120 kilo volt (kV).

Reconstructions will be made from the raw material. In addition to axial and coronal reconstructions, images series will be reconstructed in an oblique coronal image plane.

The physicist will contribute to achieve the best possible protocol. As an example it is possible to use different kV values while keeping the dose parameters (CTDIw) on the same level as for the existing temporal bone protocol. By allowing the mAs value to change, we will be able to decide on the optimal kV level for this study, without exposing some of the patients to higher radiation dose.

The physicist will also be involved in the optimisation of the reconstruction of the images of ET. The images will be reconstructed with different filters and degrees of iterative reconstruction. Using radiologists as observers, the optimal reconstruction settings for the Eustachian tube will be selected. The physicist will also calculate organ doses and effective dose for the patients.

All patients included in the study will be treated with balloon dilation in general anaesthesia, 3 - 4 weeks after the CT procedure. The ENT surgeon will be blinded to the result from the contrast media part of the CT examination. In relation to the hospital stay for balloon dilation patients will be repeatedly examined and interviewed similarly to the examination at inclusion.

Follow-up is conducted 3 months and 6 months after balloon dilatation with renewed clinical examination and interview, according to the presently established routine follow-up.

Parameters to be noted from the different time points are CT findings including contrast media passage, clinical and biochemical signs on inflammation and/or infection, symptoms related to middle ear or temporal bone disease and/or general infection, and clinical result from ET balloon dilation finally dividing the patient group into responders or non-responders from dilation.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years old Referred to ENT clinic at Rikshospitalet for evaluation and treatment of OME, tympanic membrane peroration or tympanic membrane retraction Dysfunction of the ET is suspected by the ENT surgeon The patient is a candidate for balloon dilation of the ET

Exclusion Criteria:

Previous serious allergic reaction to iodine based contrast medium Increased risk of bleeding Serious heart disease Diabetes I Previous ENT-surgery (t-tubes excluded) Middle ear disease, which requires other type of treatment Chronic rhino sinusitis or nasal polyposis Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10-20 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Extent of contrast medium passage through the Eustachian tube | 10 minutes after contrast medium application
  CT-imaging to assess contrast enhancement of the ET or pharyngeal space. Either of four alternatives is possible:
  1. Contrast enhancement of the pharyngeal space.
  2. Contrast enhancement of the ET on the oral side of the isthmus
  3. Contrast enhancement of the bony part of the ET, but not passed the isthmus
  4. No contrast enhancement of the ET

SECONDARY OUTCOMES:
Local side effects of contrast medium application | 4 weeks
  Clinical inspection
Local side effects of contrast medium application | 4 weeks
  QOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jens Petter Berg, MD, PhD, Study Director — Oslo University Hospital
Locations (1):
- Oslo UH, Oslo, Norway